CLINICAL TRIAL: NCT02742896
Title: Evaluation for Restoration of Erectile Dysfunction After Cardioversion Treatment Trial
Status: Withdrawn | Type: Observational
Sponsor: Yong Seog Oh (Other)
Responsible Party: Sponsor-Investigator, Yong Seog Oh, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: ERECT
Record Dates: First submitted 2014-10-05; First posted 2016-04-19 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; cognitive function
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Restoration of Erectile dysfunction: The changes of erectile function by using official questionnaire-The International Index of Erectile Function (IIEF)-5 1 year after conversion to sinus rhythm.
  Interventions: Other: Erectile dysfunction

INTERVENTIONS:
Other: Erectile dysfunction — The changes of erectile function by using official questionnaire-The International Index of Erectile Function (IIEF)-5 1 year after conversion to sinus rhythm.
  The changes of cognitive function by using validated assessment form-The Montreal Cognitive assessment (MoCA) 1 year after conversion to sinus rhythm.
  Other Names: official questionnaire

SUMMARY:
Erectile and Cognitive function by using the questionnaire and assessment form before sinus conversion

DETAILED DESCRIPTION:
Sinus conversion by electrical cardioversion increase cardiac output and systemic perfusion. According to recent reports, maintenance of sinus rhythm increase systemic perfusion which leads to improve renal function. Therefore, we hypothesized that sinus conversion of patients with atrial fibrillation will increase systemic perfusion which might improve the erectile dysfunction and cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to electrical cardioversion

Exclusion Criteria:

* Patients have taken any medication for erectile dysfunction or who have got any operation already or are scheduled to do.
* More than moderate degree of cognitive dysfunction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are scheduled to rhythm control of persistent atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2019-04-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
The changes of erectile function | Erectile dysfunction 1 year after conversion to sinus rhythm.
  The changes of erectile function by using official questionnaire-The International Index of Erectile Function (IIEF)-5 1 year after conversion to sinus rhythm.

SECONDARY OUTCOMES:
The changes of cognitive function | cognitive dysfunction 1 year after conversion to sinus rhythm
  The changes of cognitive function by using validated assessment form-The Montreal Cognitive Assessement(MoCA) 1 year after conversion to sinus rhythm

CONTACTS AND LOCATIONS:
Overall Officials: Yong Seog Oh, MD, Principal Investigator — Seoul St Mary hospital
Locations (1):
- Seoul St Mary's Hospital, Seoul, Seo Ch-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided